CLINICAL TRIAL: NCT03123718
Title: Prospective, Multicenter, Randomized ,Open-labeled, Phase III Study Comparing High-dose Intravenous Methotrexate Versus Intrathecal Methotrexate for the Prophylaxis of Central Nervous System Relapse in Diffuse Large B Cell Lymphoma
Brief Title: High-dose Intravenous Methotrexate Versus Intrathecal Methotrexate for Central Nervous System Prophylaxis in DLBCL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chonnam National University Hospital (Other)
Collaborators: Consortium for Improving Survival of Lymphoma (Other)
Responsible Party: Principal Investigator, Deok-Hwan Yang, Principal Investigator, Chonnam National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HDMTX
Record Dates: First submitted 2017-04-18; First posted 2017-04-21 (Actual); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: DLBCL
Keywords: methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intrathecal Methotrexate (Other)
  Interventions: Drug: Intrathecal methotrexate
- High-dose Intravenous Methotrexate (Active Comparator)
  Interventions: Drug: High-dose intravenous methotrexate

INTERVENTIONS:
Drug: Intrathecal methotrexate — Intrathecal administration of 2nd, 3rd, and 4th doses of methotrexate 15 mg and hydrocortisone 50mg on day 2 or 3 of 2nd, 3rd, and 4th cycles of immunochemotherapy with rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone (RCHOP), respectively.
  Arms: Intrathecal Methotrexate
Drug: High-dose intravenous methotrexate — Intravenous administration of 1st and 2nd doses of methotrexate 3g/m2 on day 15 of 2nd and 6th cycles of immunochemotherapy with rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone (RCHOP), respectively.
  * Dose of intravenous methotrexate will be reduced to 2g/m2 for patients aged >70 years.
  Arms: High-dose Intravenous Methotrexate

SUMMARY:
The outcome of patients with central nervous system (CNS) relapse in DLBCL is poor, with median survival times of 2-5 months. This fatal prognosis necessitates CNS prevention in a subgroup of patients with a high risk of CNS relapse.

Intrathecal methotrexate (ITMTX) has traditionally been used, although its efficacy for CNS prophylaxis is contradictory. High-dose intravenous methotrexate (IVMTX) has been suggested as an alternative approach. Considering the lack of evidence supporting the role of ITMTX, the investigators propose to compare the efficacy of ITMTX and IVMTX for prophylaxis of CNS relapse in a subgroup of patients with DLBCL at a high risk for CNS relapse.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years <80
* Newly diagnosed, histologically confirmed DLBCL
* High-risk of CNS recurrence at diagnosis:

  1. Age-adjusted IPI (aaIPI) ≥2 or IPI ≥4 with extranodal involvement of >1 site plus serum lactate dehydrogenase (LDH) > normal OR
  2. Involvement of high-risk locations: bone marrow, nasal or paranasal sinuses, testis, epidural disease (paravertebral or vertebra), breast, adrenal or kidney
* Estimated life expectancy of more than 90 days
* Performance status (ECOG) ≤ 2
* Written informed consent

Exclusion Criteria:

* Psychiatric or mental disorder which make the patient unable to give an informed consent and/or adhere to the protocol
* DLBCL or following subtypes:

  1. Primary mediastinal large B-cell lymphoma
  2. Grey zone lymphoma)
  3. Primary cutaneous DLBCL
* Previous immunochemotherapeutic treatment for DLBCL other than short-term use of corticosteroids (≤ 8 days before randomization)
* Previous radiotherapy
* CNS involvement of DLBCL at diagnosis
* HIV positive
* Any contraindication for application of RCHOP or high dose methotrexate
* Any of following laboratory results

  1. Absolute neutrophil count < 1,500 cells/mm3 (1.5 x 109/L),
  2. Platelet count < 100,000/mm3 (100 x 109/L), or < 75,000 /mm3 in patients with bone marrow involvement,
  3. Serum aspartate transaminase or serum alanine transaminase ≥3.0 x upper limit of normal (ULN),
  4. Serum total bilirubin > 2 x ULN (with the exception of hemolytic anemia),
* Serum creatinine >2.0 x ULN or creatinine clearance <50 mL/min
* Active cancer except curable basal cell carcinoma, cervical cancer in situ, and/or papillary thyroid cancer during the last five years
* Ejection fraction < 45% on echocardiography
* Uncontrolled active hepatitis
* Pregnancy or breast-feeding
* Men and women of reproductive potential no agreeing to use an acceptable method of birth control during treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of CNS relapse | 2 year
  The rate of relapse will be analyzed by the cumulative incidence method

SECONDARY OUTCOMES:
Toxicity | 2 year
  Toxicity will be graded according to NCI-CTCAE v.4.03
Progression-free survival (PFS) | 2 year
  PFS will be calculated from randomization to the date of CNS relapse and/or systemic disease progression, death, or last follow-up, as appropriate.

CONTACTS AND LOCATIONS:
Locations (1):
- Chonnam National University Hwasun Hospital, Hwasun-gun, Jeollanam-do, South Korea

IPD SHARING:
Plan to Share IPD: No